CLINICAL TRIAL: NCT03776721
Title: Treatment of Breast Cancer-related Lymphedema With Stem Cells and Fat Grafting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Mads Gustaf Jørgensen, Principal Investigator, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S-20180117
Record Dates: First submitted 2018-11-12; First posted 2018-12-17 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema | interventions — Lipectomy; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All patients undergo the same liposuction procedure. During general anesthesia, patients are randomized to either fat grafting or sham grafting with saline injection to the axilla. After stem cell suspension, patients receive either stem cell or saline injection depending on randomization using masked syringes.
  Participants are blinded, care providers postoperatively are blinded, primary investigator is blinded and all outcome assessors are blinded. The surgeon performing the liposuction and the stem-cell staff are unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active treatment (Experimental)
  Interventions: Procedure: Liposuction; Procedure: Fat graft; Biological: Stem cell injection
- Placebo treatment (Placebo Comparator)
  Interventions: Procedure: Liposuction; Procedure: Sham graf (Saline injection); Procedure: Saline injection

INTERVENTIONS:
Procedure: Liposuction — Liposuction is performed on the abdomen or thighs.
Procedure: Fat graft — 30mL harvested lipoaspirate is injected at the affected axillary site.
  Other Names: lipotransfer
  Arms: Active treatment
Procedure: Sham graf (Saline injection) — 30mL saline is injected at the affected axillary site.
  Arms: Placebo treatment
Biological: Stem cell injection — 4mL stem cell suspension injected at the affected axillary site.
  Arms: Active treatment
Procedure: Saline injection — 4mL saline injected at the affected axillary site.
  Arms: Placebo treatment

SUMMARY:
Breast cancer-related lymphedema is one of the most common and feared consequences of breast cancer treatment. Currently, lymphedema is primarily addressed conservatively with compression garments. Regenerative medicine may provide a new treatment option for lymphedema. This Phase 3 trial will examine the efficacy, effectiveness and safety of freshly isolated adipose-derived stromal cells administered in conjunction with a fat grafting procedure to the affected axillary region.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral arm lymphedema secondary to breast cancer treatment including lymph node dissection.
* Cancer free for at least 1 year
* The patient understands the nature and purpose of this study and the study procedures and has signed informed consent.
* The opposite upper extremity is healthy (no lymphedema).
* ASA score of 1 or 2.
* The patient is able to read, understand, and complete Danish questionnaires.
* Pitting lymphedema ISL grade 1 or 2.
* A minimum circumference difference of 2cm or a minimum volume difference of 200mL.

Exclusion Criteria:

* Pregnant or lactating.
* Bilateral lymphedema
* Current or previous malignancies other than breast cancer.
* Insulin-dependent diabetes.
* Diagnosed with any form of psychotic disorder, which may impact study participation.
* Not ceased smoking during treatment.
* Active implantables (e.g. pacemaker or neurostimulator)
* Unrealistic treatment expectations.
* Known hepatitis, HIV or syphilis infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Change in arm volume | Baseline, 3, 6, 9 and 12 months
  Assessed using clinical circumference measurement

SECONDARY OUTCOMES:
Safety of treatments: Assessed by asking the patient at each visit | Baseline, 3, 6, 9 and 12 months
  Any side effects to treatments. Assessed by asking the patient at each visit.
Subjective changes assessed using the LYMPH-ICF (Lymphoedema Functioning, Disability and Health) questionaire | Baseline, 3, 6, 9 and 12 months
  Subjective change of lymphedema assessed by questionnaire. Range: 0-100. 100 being the most bothered.
Subjective changes assessed using DASH (DISABILITIES OF THE ARM, SHOULDER AND HAND) questionaire | Baseline, 3, 6, 9 and 12 months
  Subjective change of lymphedema assessed by questionnaire. Range: 1-5. 5 being the most bothered
Subjective changes assessed using SF-36 questionnaire | Baseline, 3, 6, 9 and 12 months
  Subjective change of quality of life assessed by questionnaire. Range: 0-100. 0 being the most bothered.
Change in lymph drainage | Baseline and 12 months
  Change in lymph drainage assessed by indocyanine-green lymphangiography
Change in conservative lymphedema treatment | Baseline, 3, 6, 9 and 12 months
  Change in use or type of conservative lymphedema treatments
Change in adverse lymphedema-related events | Baseline, 3, 6, 9 and 12 months
  Change in infection rates and sick-days due to lymphedema.
Change in L-DEX score (bioimpedance) | Baseline, 3, 6, 9 and 12 months
  Change in L-DEX score of lymphedema arm derived from bioimpedance. Higher values mean more fluid in the lymphedema arm compared to the healthy arm.
Change in weight and arm tissue composition | Baseline, 3, 6, 9 and 12 months
  Assessed using dual energy x-ray absorptiometry (DXA) scan. Change in values from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jens A Sørensen, MD, PhD, Study Chair — Department of Plastic Surgery, Odense University Hospital
Locations (1):
- Department of Plastic and Reconstructive Surgery, Odense, Denmark

REFERENCES:
- [Derived] Jorgensen MG, Jensen CH, Hermann AP, Andersen DC, Toyserkani NM, Sheikh SP, Sorensen JA. No Clinical Efficacy of Adipose-Derived Regenerative Cells and Lipotransfer in Breast Cancer-Related Lymphedema: A Double-Blind Placebo-Controlled Phase II Trial. Plast Reconstr Surg. 2024 Dec 1;154(6):1172-1182. doi: 10.1097/PRS.0000000000011343. Epub 2024 Feb 7. PMID 39591365